CLINICAL TRIAL: NCT02302989
Title: Prospective Double-blind Randomized Study to Evaluate Lucentis for Prophylaxis Against the Conversion to Neovascular Age-related Macular Degeneration (AMD) in High-risk Eyes (Let's ProTECT AMD Eyes)
Brief Title: Prophylactic Ranibizumab for Exudative Age-Related Macular Degeneration
Acronym: PROTECT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leonard Feiner, MD, PhD (Other)
Collaborators: NJ Retina (Retina Associates of New Jersey) (Other)
Responsible Party: Sponsor-Investigator, Leonard Feiner, MD, PhD, Principal Investigator, NJ Retina (Retina Associates of New Jersey)
Organization: NJ Retina (Retina Associates of New Jersey) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ML29346
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): No treatment. Observation only
- Quarterly Ranibizumab 0.5 (Active Comparator): Quarterly intravitreal injection of 0.5mg Ranibizumab Intervention: Drug: Ranibizumab 0.5mg
  Interventions: Drug: Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Ranibizumab 0.5mg
  Other Names: Lucentis
  Arms: Quarterly Ranibizumab 0.5

SUMMARY:
To evaluate Ranibizumab as prophylaxis against the conversion to neovascular Age-Related Macular Degeneration

DETAILED DESCRIPTION:
This is an open-label, prospective, randomized study of intravitreally administered ranibizumab 0.5 mg in subjects with unilateral neovascular AMD in which the fellow (study) eye is at high-risk for also developing conversion to neovascular AMD.

The Study will determine the efficacy of a quarterly injection of Ranibizumab to prevent the conversion of dry age-related macular degeneration to neovascular AMD in high risk eyes.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50 years old
* Able to sign informed consent and comply with the study protocol for the duration of the two years.
* Nonexudative age-related macular degeneration (AMD) in one eye (study eye) •At time of enrollment, fellow non-study eye must have recently diagnosed (not more than 2 years prior to enrollment), angiographically documented, previously untreated prior to diagnosis, CNV lesion (i.e., leakage on fluorescein angiography AND subretinal, intraretinal, or sub-RPE fluid on OCT) secondary to age-related macular degeneration.

Exclusion Criteria:

* Previous treatment with verteporfin PDT, Macugen®, Lucentis®, intravitreal Avastin®, intravitreal Eylea®, thermal laser, external beam radiation or other AMD therapy in the study eye.
* History of macular hole in study eye.
* History of vitrectomy in study eye.
* Lens extraction or implantation within the last 3 months.
* Capsulotomy within the last 1 month.
* Lens or other media opacity that would preclude good fundus photography or angiography within the next 2 years.
* Nevus > 2 disc areas within 3000 microns of the foveal center or with fluid or leakage on fluorescein angiography.
* Macular edema or signs of diabetic retinopathy more severe than 10 red dots (microaneurysms or blot hemorrhages).
* Retinal changes related to high myopia and no myopic correction greater than 8.00 diopters spherical equivalent [sphere + ½ cylinder].
* Any progressive ocular disease that would affect visual acuity within the next 2 years.
* Previous participation in any studies of investigational drugs likely to have ocular effects within 30 days preceding the initial study treatment.
* Concurrent use of systemic anti-VEGF agents.
* Active or recent (within 4 weeks) intraocular inflammation (grade trace or above) in the study eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* For subjects who have undergone prior refractive or cataract surgery in the study eye, the preoperative refractive error in the study eye cannot exceed 8 diopters of myopia.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure > 25 mmHg) despite treatment with antiglaucoma medication).
* Patients who are unable to be photographed to document CNV due to known allergy to fluorescein dye, lack of venous access or cataract obscuring the CNV.
* Patients with other ocular diseases that can compromise the visual acuity of the study eye such as amblyopia and anterior ischemic optic neuropathy.
* Current treatment for active systemic infection.
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders.
* History of recurrent significant infections or bacterial infections.
* Inability to comply with study or follow-up procedures.
* Pregnancy (positive pregnancy test) or lactation Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Conversion to neovascular AMD. (CNV leakage on FA and evidence of any fluid on SD-OCT) | 2 years
  The development of CNV will be assessed by CNV leakage on FA and evidence of any fluid on SD-OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Feiner, MD, MD, PhD, Principal Investigator — NJ Retina (Retina Associates of New Jersey)
Locations (2):
- United States (2):
  - NJ Retina (Retina Associates of New Jersey), Teaneck, New Jersey
  - NJ Retina (Retina Associates of New Jersey), Vauxhall, New Jersey